CLINICAL TRIAL: NCT01222468
Title: A Randomized Double-Blinded Crossover Trial Assessing the Effect of Cannabinoids on Spasticity and Neuropathic Pain in Spinal Cord Injured Persons
Brief Title: Effect of Cannabinoids on Spasticity and Neuropathic Pain in Spinal Cord Injured Persons
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: The Manitoba Spinal Cord Injury Research Fund (Unknown); Canadian Paraplegic Association (Other); Health Sciences Centre Foundation, Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Karen Ethans, Principal Investigator MD, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1976
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Muscle Spasticity as a Result of Spinal Cord Injury
Keywords: Spasticity, Spinal Cord Injury
MeSH Terms: conditions — Muscle Spasticity; Spinal Cord Injuries | interventions — nabilone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- nabilone (Active Comparator): nabilone 0.5 mg tablets dose-titrated over an 11-week period to a maximum of 3mg po daily. Subjects are allowed to drop back to the previous dose following a dose increase once if required
  Interventions: Drug: nabilone 0.5 mg
- placebo (Placebo Comparator): look-alike 0.5 mg placebo tablets titrated to a maximum daily dose of 3.0 mg daily over an 11-week phase. Subjects are allowed to drop back to the previous dose following a dose increase once during the 11-week phase if required
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: nabilone 0.5 mg — nabilone 0.5 mg tablets od titrated to a maximum daily dose of 3mg po over an 11-week phase
  Other Names: Cesamet
  Arms: nabilone
Drug: placebo — placebo 0.5 mg po daily, dose titrated to a maximum daily dose of 3.0mg po over an 11-week phase
  Arms: placebo

SUMMARY:
This study is being conducted to study the effect of nabilone (a synthetic cannabinoid)on spasticity in spinal cord injured persons.The study will be a phase 2, randomized, placebo-controlled crossover study. Each eligible subject will participate for 26 weeks.Subjects will be randomized to receive either nabilone or placebo during phase 1 of the study. Study drug will be titrated up from 0.5mg daily to a maximum of 3.0 mg daily over the first 11-week phase. Following a 4-week washout period, subjects will be crossed-over to the opposite arm for another 11 week treatment period (phase 2).

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury
* 12 months post -injury
* C2-T12, ASIA A-D, stable level of injury
* moderate to severe spasticity or moderate to severe neuropathic pain
* no cognitive impairment
* spasticity medications unchanged for at least 30 days or inadequate pain control at a stabilized dose of either gabapentin or pregabalin for at least 30 days
* no botulinum toxin injections x 6 months

Exclusion Criteria:

* significant cardiovascular disease
* major illness in another body area
* history of psychological disorders or predisposition to psychosis
* sensitivity to cannabinoids
* severe liver disfunction
* history of drug dependancy
* fixed tendon contractures
* used cannabis in the past 30 days
* unwilling to refrain from smoking cannabis during the study
* pregnant or nursing mother

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Ashworth Scale | 26 weeks
  A scale that grades resistance to rapid passive movement across a relaxed joint on an ordinal scale of 0 to 4.
VAS (visual analog scale)pain intensity scale | 26 weeks
  Primary outcome measure for pain will be a change in the VAS pain intensity scale. Using a visual intensity scale, patients are asked to record their daily pain score over the previous 24 hours.

SECONDARY OUTCOMES:
Sum of the Ashworth Scale in the eight muscle groups of each side of the body. | 26 weeks
  As above
Penn Spasm Frequency Scale | 26 weeks
  Scale graded by study participants to measure frequency of muscle spasms throughout the period in question
Visual Analog Scale | 26 weeks
  Patients rate the intensity of their spasms on a 100 mm pencil and paper VAS scale
Pittsburgh Sleep Quality Index | 26 weeks
  Questionnaire that measures patient-reported sleep quality that will be administered at Visits 1,6 and 12
Subject's Global Impression of Change | 26 weeks
  Questionnaire that asks the subject to rate his or her impression of the effects of the study medication.
Clinician's Global Impression of Change | 26 weeks
  Questionnaire that asks the Clinician to rate his or her impression of the effect of study medication.
VAS Pain Impact Scale | 26 weeks
  A continuous scale measuring the impact of pain with 0mm being non-disruptive and 100 mm being incapacitating
The Short Form McGill Pain Questionnaire (SF-MPQ) | 26 weeks
  A questionnaire with 3 components: a VAS to determine overall pain levels, a 15-word list of pain descriptors; and a Present Pain Intensity Scale to determine patient's pain at the time of survey completion
Neuropathic Pain Questionnaire | 26 weeks
  A clinician-administered questionnaire consisting of both sensory descriptors and signs related to bedside sensory examination

CONTACTS AND LOCATIONS:
Overall Officials: Karen D. Ethans, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre Rehabilitation Hospital, Winnipeg, Manitoba, Canada